CLINICAL TRIAL: NCT07381660
Title: Stereotactic Body Radiotherapy (SBRT) Versus Surgical Resection in Patients With Small Hepatocellular Carcinoma: A Phase III, Open-label, Randomized Controlled Trial
Brief Title: SBRT Versus Surgical Resection for Small HCC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Chen Min-Shan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2025-806-01
Record Dates: First submitted 2026-01-16; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: HCC; SBRT; Resection
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resection (Active Comparator): Patient receive surgical resection
  Interventions: Procedure: Resection
- SBRT (Experimental): Patient receive SBRT
  Interventions: Radiation: Stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy (SBRT) — The SBRT dose ranges from 33 to 54 Gy and is delivered in three fractions on alternate days, with treatment completed within one week. This study enrolls patients with small hepatocellular carcinoma, defined as a solitary tumor with a maximum diameter of ≤5 cm, and compares the efficacy of SBRT with that of surgical resection.
  Arms: SBRT
Procedure: Resection — Surgical resection serves as the control treatment in this study
  Arms: Resection

SUMMARY:
Hepatocellular carcinoma (HCC) is one of the leading causes of cancer-related incidence and mortality in China and represents a major public health challenge. Surgical resection is the most commonly used curative treatment for HCC and can provide favorable long-term outcomes. However, resection is associated with substantial perioperative morbidity, and its applicability is limited in certain patient populations, including those with recurrent disease, those who have undergone conversion therapy, and those with significant coexisting medical conditions.

Advances in radiotherapy technology and the development of highly precise delivery techniques have led to the increasing use of stereotactic body radiotherapy (SBRT) in the management of HCC, particularly in patients with small tumors. Randomized controlled trials conducted by our group have shown that, in patients with recurrent small HCC, SBRT provides superior local tumor control compared with radiofrequency ablation. These findings suggest that SBRT may represent a potentially curative treatment option for selected patients with small HCC.

On the basis of this evidence, the present study is designed to compare the efficacy and safety of surgical resection and SBRT in patients with small HCC. Patients with a solitary tumor measuring 5 cm or less in maximum diameter will be randomly assigned to undergo either surgical resection or SBRT. The primary end point of the study is overall survival. This trial aims to define the relative benefits and risks of these two treatment strategies and to provide high-quality evidence to inform clinical decision making and future guideline recommendations.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 75 years, with no restriction on sex;
2. Clinically or pathologically diagnosed hepatocellular carcinoma, according to the Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2024 edition);
3. A solitary tumor with a maximum diameter of ≤5 cm, for which treatment is indicated;
4. No radiologic evidence of macrovascular invasion, distant metastasis, or lymph node metastasis;
5. Treatment-naïve or previously treated patients are eligible, provided that they are deemed suitable for both surgical resection and radiotherapy by a multidisciplinary team (MDT) and do not require concomitant systemic therapy at enrollment;
6. For patients with recurrent disease, recurrence must occur at least 1 year after prior curative treatments;
7. Previously treated patients must not have received systemic therapy within 6 months before enrollment;
8. In previously treated patients, tumor size must be assessed according to RECIST version 1.1 at enrollment;
9. A normal liver volume of ≥700 cc, with an estimated future liver remnant volume of >40% after resection;
10. A Karnofsky performance-status score of ≥90;
11. Child-Pugh class A liver function;
12. An estimated life expectancy of more than 6 months;
13. Adequate organ function, defined as follows: white-cell count ≥3.5×10⁹/L, absolute neutrophil count ≥1.5×10⁹/L, platelet count ≥75.0×10⁹/L, hemoglobin ≥90 g/L; serum albumin ≥28 g/L; total bilirubin ≤1.5 times the upper limit of normal (ULN), alanine aminotransferase or aspartate aminotransferase ≤2.5 times the ULN; serum creatinine ≤1.5 times the ULN or creatinine clearance >60 mL per minute; and no severe concomitant organic disease;
14. The ability to understand the study procedures and to provide written informed consent before the initiation of any study-specific procedures, with agreement to receive treatment and follow-up according to the study protocol.

Exclusion Criteria:

1. Severe dysfunction of major organs, including the heart, lungs, or kidneys; active infection other than viral hepatitis; or other serious concomitant conditions that preclude tolerance of either surgery or radiotherapy;
2. Contraindications to surgical resection or radiotherapy;
3. A history of other malignant tumors, with the exception of nonmelanoma skin cancer, carcinoma in situ of the cervix, or previously cured prostate cancer, nasopharyngeal carcinoma, breast cancer, or early-stage laryngeal cancer;
4. A history of multiple abdominal surgeries or liver or other solid-organ transplantation;
5. Previous radiotherapy to the upper abdomen;
6. Pregnancy or breastfeeding;
7. Any other condition that may interfere with patient enrollment or the assessment of study outcomes;
8. Refusal to comply with the follow-up requirements of the study protocol or refusal to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
OS | time from random assignment to death from any cause, assessed up to 100 months
  time from random assignment to death from any cause

SECONDARY OUTCOMES:
PFS | time from random assignment to tumor progression or death fromany cause, assessed up to 100 months
  time from random assignment to tumor progression or death fromany cause
LPFS | time from random assignment to local tumor progression or death fromany cause, assessed up to 100 months
  time from random assignment to local tumor progression or death fromany cause

IPD SHARING:
Plan to Share IPD: Yes
IPD are available from the corresponding author (Minshan Chen and Yaojun Zhang) by request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months and ending 2 years after the publication of results
Access Criteria: For academic discussion purposes, investigators who are interested in this study may contact the study team by email to request the study protocol, the statistical analysis plan, and other relevant materials.
URL: https://www.researchdata.org.cn/